CLINICAL TRIAL: NCT05019508
Title: Fetal Cardiac Function Parameters and HbA1c As Screening for Gestational Diabetes Mellitus: a Pilot Study
Brief Title: Fetal Cardiac Function Parameters and HbA1c As Screening for Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Christopher S. Ennen, Associate Professor of Medicine, University of Virginia
Other Study IDs: 210175
Record Dates: First submitted 2021-08-09; First posted 2021-08-25 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2023-08

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- High Risk for Gestational Diabetes Mellitus (GDM): High risk women screened with HbA1c at initiation of prenatal care who were not diagnosed with Type 2 Diabetes Mellitus or Early GDM.
  These women will have Fetal Cardiac Function Parameters at their 20 week anatomy scan (E/A ratio, IVS, MPI). At their 24-28 week routine GDM screening, we will repeat the HbA1c and will repeat the E/A ratio, IVS, MPI. If women have a growth scan for any reason between 32 and 36 weeks, E/A ratio, IVS, and MPI will be repeated at those times.

SUMMARY:
This is a prospective cohort study to assess the predictive value of fetal cardiac parameters, the change in fetal cardiac parameters (CFP), HbA1c, and/or the change in HbA1c (ΔHbA1c) for gestational diabetes.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is the onset of carbohydrate intolerance that affects up to 6-9% of pregnancies. A diagnosis of GDM conveys numerous implications for the health of the mother and the fetus if not properly identified and/or treated. Maternal complications include increased risk of preeclampsia and development of Type 2 diabetes mellitus later in life. The risks to the fetus include increased risk of macrosomia, stillbirth, hypoglycemia, shoulder dystocia as well as increased risk of childhood obesity and diabetes.

Per ACOG guidelines, women who are at an increased risk for undiagnosed pre-gestational diabetes mellitus or developing GDM should receive early screening when they initially present for prenatal care, most commonly in the late first or early second trimester.5 The best test for this early assessment is not yet established. Practices patterns vary between use of the two-step oral glucose tolerance screening and glycated hemoglobin (HbA1c). Use of the oral glucose tolerance tests for screening of GDM is well-established and the cut-offs determined for 24-28 week routine screening are used when the oral tolerance tests are administered in early pregnancy. An HbA1c level ≥6.5% is used to diagnose diabetes, however there is evidence that there is a higher rate of GDM diagnosis and poor outcomes with a HbA1c level as low as 5.6%. Women who are not diagnosed with GDM before 20 weeks, go on to routine screening at 24-28 weeks.

With the current protocols for early GDM screening, treatment of early glucose intolerance has not shown to improve neonatal outcomes, however. The methods and timing of current early GDM screening may not be identifying a population that is truly at risk of poor outcomes from glucose intolerance in the way routine screening with the two-step process does. More research into screening paradigms other than oral tolerance tests in early pregnancy is needed. A HbA1c level assesses the amount glycation of hemoglobin molecules in red blood cells, indirectly estimating the average blood glucose level over the past 8-12 weeks. HbA1c independently has not been shown to be adequately predictive of a GDM diagnosis in pregnancy. Many studies assessing the screening value of HbA1c obtain the value in the first trimester when a large portion of the 12 weeks prior is before significant placentation. A change in HbA1c in the first half of pregnancy, when combined with other clinical variables may be more predictive. Novel clinical variables should also be considered. There is evidence that even well-control pre-gestational and gestational diabetics show significant variation in fetal cardiac functional parameters such as interventricular septum thickness (IVS), the E/A ratio, and myocardial performance index (MPI). The predictive value of these changes for glucose intolerance has not yet been investigated.

This is be a prospective cohort study to assess the predictive value of fetal cardiac parameters, the change in fetal cardiac parameters (CFP), HbA1c, and/or the change in HbA1c (ΔHbA1c) for gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who have completed a HbA1c test during the first 20 weeks of pregnancy.
* Risk for GDM including any of the following:

  * Obese
  * History of GDM
  * History of macrosomia
  * Twin gestation
  * PCOS
  * Family history of diabetes

Exclusion Criteria:

* • Pregnant women who have not completed a HbA1c test during the first 20 weeks of pregnancy.

  * women with pre-gestational diabetes
  * nonviable pregnancy
  * fetal anomalies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All pregnant women being see in the Maternal Fetal Medicine clinic at the Battle Building at the University of Virginia.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
We will assess the predictive ability of fetal Cardiac Function Parameter for diagnosis of Gestational Diabetes Mellitus by oral glucose tolerance tests | one year
  Area under the curve statistics will be used to assess values of CFP, ΔCFP, ΔHbA1c (independently and in conjunction) which maximize sensitivity, specificity, and PPV for GDM.

SECONDARY OUTCOMES:
Secondary outcomes | one year
  Secondary outcomes will be the change in fetal cardiac function parameters (ΔCFP) between 20 weeks and 24-28 weeks assessments, HbA1c results, ΔHbA1c results, diagnosis of GDM.
Secondary neonatal outcomes | one year
  These include birth weight, hypoglycemia, NICU admission etc.

CONTACTS AND LOCATIONS:
Overall Officials: Christoher Ennen, MD, Study Director — UVA
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States